CLINICAL TRIAL: NCT00609271
Title: Macronutrient Composition of Diet and Risk Factors for Cardiovascular Disease
Brief Title: Study of Macronutrients and Heart Disease Risk
Acronym: MACRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Lydia A. Bazzano, Associate Professor Epidemiology, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-00111
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Body Composition; Blood Pressure; Cardiovascular Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): low carbohydrate diet
  Interventions: Behavioral: low carbohydrate diet
- 2 (Active Comparator): low fat diet
  Interventions: Behavioral: low fat diet

INTERVENTIONS:
Behavioral: low carbohydrate diet — <40 grams carbohydrate/day
  Arms: 1
Behavioral: low fat diet — <30% fat, <7% saturated fat
  Arms: 2

SUMMARY:
The objective of this trial is to examine the long-term effects of a diet low in carbohydrates, as compared to one low in fat, on cardiovascular disease risk factors, including blood pressure (BP), body weight and composition, serum lipids, plasma glucose, insulin, adipocytokines (adiponectin, leptin, resistin), and C-reactive protein (CRP) among obese adults.

The investigators will test the following hypotheses:

Hypothesis 1: Compared to a low fat diet, a diet low in carbohydrates will reduce systolic and diastolic BP over 12 months; Hypothesis 2: Compared to a low fat diet, a diet low in carbohydrates will reduce body weight, total percent body fat, and waist circumference over 12 months; Hypothesis 3: Compared to a low fat diet, a diet low in carbohydrates will reduce serum levels of LDL-cholesterol and triglycerides and increase serum levels of HDL-cholesterol over 12 months; Hypothesis 4: Compared to a low fat diet, a diet low in carbohydrates will reduce plasma levels of glucose and insulin levels over 12 months; and Hypothesis 5: Compared to a low fat diet, a diet low in carbohydrates will reduce plasma levels of leptin, resistin, and CRP and increase plasma levels of adiponectin over 12 months.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) remain the leading cause of death globally as well as here in the United States. Manipulations of the macronutrient (protein, carbohydrate and fat) contents of diet have been used extensively for weight loss and weight control in the past several decades. Low carbohydrate diets, in particular, have gained popularity for weight loss. However, few studies have examined the effects of a diet low in carbohydrates on traditional and novel cardiovascular risk factors in the long term, particularly in contrast to the current dietary recommendations for decreased fat intake to reduce risk of CVD. In this proposal, we plan to conduct a 12-month, parallel-arm, randomized controlled trial of a diet low in carbohydrates versus the currently recommended low fat diet to reduce CVD risk factors among obese adults. The objective of this trial is to examine the long-term effects of a diet low in carbohydrates, as compared to one low in fat, on CVD risk factors, including blood pressure (BP), body weight and composition, serum lipids, plasma glucose, insulin, adipocytokines (adiponectin, leptin, resistin), and C-reactive protein (CRP) among obese adults. In order to accomplish these objectives we will randomize 130 eligible participants (n=65 in each group) to consume either a diet low in carbohydrates (≤40 g/d) or a diet low in fat (<7% saturated fat, <30% total fat). Neither of the diets will be energy-restricted. Participants will meet with a dietitian for one-on-one counseling sessions weekly for the first 4 weeks, then bi-monthly in small group sessions for the next 5 months, and monthly in larger group sessions for the final 6 months of the intervention. Data on both traditional and novel CVD risk factors will be collected at baseline, 3, 6, and 12 months. We hypothesize that a diet low in carbohydrates as compared to a diet low in fat will lower systolic and diastolic BP, body weight, total percent body fat, waist circumference, serum levels of triglycerides, and plasma levels of insulin, glucose, leptin, resistin, and CRP, and increase serum levels of HDL-cholesterol and adiponectin. Because CVD is the most common cause of death here in the U.S. and world-wide, this study has important public health implications. It will provide new information on the potential long-term effects of diets low in carbohydrates on both the traditional risk factors for CVD as well as novel risk factors and inflammatory factors. The results from this study will help to determine if a diet low in carbohydrates as compared to the currently recommended low fat diet can decrease the risk of CVD among obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 22 - 75 years, any race/ethnicity
* BMI of 30 - 45 k/m2
* Willing and able to provide informed consent

Exclusion Criteria:

* History of self-reported clinical CVD (angina/myocardial infarction, coronary revascularization, heart failure, stroke/transient ischemic attack, peripheral arterial disease)
* Medical condition in which a low-carbohydrate diet may not be advised (diabetes, renal disease, cancer requiring treatment during the past year, osteoporosis, untreated thyroid disease, gout)
* Current use of more than 2 antihypertensive or more than 2 cholesterol-lowering medications
* For women, current pregnancy or breastfeeding or plans to become pregnant during the study period
* Consumption of more than 21 alcoholic beverages per week
* Currently on a diet or using prescription weight loss medications, underwent weight loss surgery, and/or experienced weight loss >15 pounds within 6 months of study entry
* Plans to move out of the study area (>1 hour from study site) or difficulty to come to the study site
* Participation of another household member in the study; employees or persons living with employees of the study
* Participation in other lifestyle intervention trials currently
* At the discretion of the study coordinator

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia A Bazzano, MD, PhD, Principal Investigator — Tulane University
Locations (1):
- Tulane University, Office of Health Research, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Hu T, Yao L, Reynolds K, Niu T, Li S, Whelton P, He J, Bazzano L. The effects of a low-carbohydrate diet on appetite: A randomized controlled trial. Nutr Metab Cardiovasc Dis. 2016 Jun;26(6):476-88. doi: 10.1016/j.numecd.2015.11.011. Epub 2015 Dec 12. PMID 26803589
- [Derived] Bazzano LA, Hu T, Reynolds K, Yao L, Bunol C, Liu Y, Chen CS, Klag MJ, Whelton PK, He J. Effects of low-carbohydrate and low-fat diets: a randomized trial. Ann Intern Med. 2014 Sep 2;161(5):309-18. doi: 10.7326/M14-0180. PMID 25178568

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Started | 75 | 73
Completed | 59 | 60
Not Completed | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Carbohydrate Diet | Low Fat Diet | Total
Number analyzed (Participants) | 75 | 73 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (9.9) | 47.8 (10.4) | 46.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 131
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 33 | 67
  Black | 40 | 36 | 76
  Asian | 1 | 0 | 1
  Hispanic | 0 | 3 | 3
  Other | 0 | 1 | 1
body weight [Mean (Standard Deviation); unit: kg] | 96.3 (12.7) | 97.9 (13.5) | 97.1 (13.1)
body composition [Mean (Standard Deviation); unit: %]
  Fat mass | 40 (10) | 40 (10) | 40 (10)
  Lean Mass | 60 (10) | 60 (10) | 60 (10)
body mass index [Mean (Standard Deviation); unit: kg/m**2] | 35.2 (3.8) | 35.6 (4.5) | 35.4 (4.2)
waist circumference [Mean (Standard Deviation); unit: cm] | 108.4 (9.3) | 111.0 (10.7) | 109.7 (10.1)
systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 120.3 (12.8) | 124.9 (13.8) | 122.6 (13.5)
diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 77.5 (9.0) | 79.4 (8.3) | 78.4 (8.7)
total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 198.8 (42.2) | 204.3 (40.7) | 201.5 (41.5)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 122.5 (34.6) | 122.7 (38.6) | 122.6 (36.6)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 53.8 (13.3) | 56.5 (12.8) | 55.1 (13.1)
total-HDL cholesterol ratio [Mean (Standard Deviation); unit: unitless] | 3.8 (1.0) | 3.8 (1.0) | 3.8 (1)
triglycerides [Mean (Standard Deviation); unit: mg/dL] | 112.6 (54.1) | 125.5 (81.3) | 119.0 (69.1)
plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 94.5 (10.9) | 93.4 (9.2) | 94.0 (10.1)
serum insulin [Mean (Standard Deviation); unit: pmol/L] | 102.8 (63.9) | 105.6 (54.9) | 104.2 (59.7)
serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.0 (0.2) | 1.1 (0.2) | 1.0 (0.1)
C-reactive protein [Mean (Standard Deviation); unit: nmol/L] | 46.7 (40.0) | 46.7 (48.6) | 46.7 (44.5)
Medication use [Count of Participants; unit: Participants]
  Antihypertensive | 21 | 24 | 45
  Lipid-Lowering | 12 | 9 | 21
Physical activity level [Mean (Standard Deviation); unit: MET-h/wk] | 16.3 (26.0) | 19.6 (35.5) | 17.9 (31.1)
Framingham risk percent [Mean (Standard Deviation); unit: %] — The Framingham Risk score predicts the 10-year risk of developing coronary heart disease (CHD). Risk is predicted based on gender-specific tables provided by Wilson et al (Circulation 1998: 1837-47) comprised of the sum of points obtained from the following factors: age, presence of diabetes, cigarette smoking, blood pressure, high density lipoprotein level, and total cholesterol level.
  Risk calculated from this score can range from a 1% chance of developing CHD to a >= 56% chance of developing CHD in men --- and a 1% chance of developing CHD to a >=32% chance of developing CHD in women.
  % | 3.9 (3.1) | 4.2 (3.3) | 4.0 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Predicted Mean Difference in Body Weight From Baseline, by Assigned Dietary Group
Description: Predicted mean difference from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
kg
  Change in body weight after 3 months | -5.7 [-6.5 to -4.9] | -2.6 [-3.4 to -1.7]
  Change in body weight after 6 months | -5.6 [-6.5 to -4.6] | -2.3 [-3.3 to -1.3]
  Change in body weight after 12 months | -5.3 [-6.8 to -3.8] | -1.8 [-3.3 to -0.3]

2. Primary Outcome: Predicted Mean Differences in Lean Mass From Baseline, by Assigned Dietary Group
Description: Mean Difference in Lean Mass predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: % of body weight that is lean mass
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
% of body weight that is lean mass
  Change of % lean mass after 3 months | 1.6 [1.0 to 2.2] | 0.4 [-0.2 to 1.1]
  Change of % lean mass after 6 months | 1.5 [0.9 to 2.1] | 0.2 [-0.4 to 0.7]
  Change of % lean mass after 12 months | 1.3 [0.5 to 2.0] | -0.4 [-1.2 to 0.4]

3. Primary Outcome: Predicted Mean Differences in Fat Mass From Baseline, by Assigned Dietary Group
Description: Mean Difference in Fat Mass predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: % body weight that is fat mass
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
% body weight that is fat mass
  Change of % fat mass after 3 months | -1.1 [-1.7 to -.05] | -0.3 [-0.9 to 0.3]
  Change of % fat mass after 6 months | -1.1 [-1.7 to -0.6] | -0.1 [-0.6 to 0.5]
  Change of % fat mass after 12 months | -1.2 [-2.0 to -0.4] | 0.3 [-0.5 to 1.1]

4. Primary Outcome: Predicted Mean Differences of Waist Circumference From Baseline, by Assigned Dietary Group
Description: Predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
cm
  Change in waist circumference after 3 mo | -5.5 [-6.6 to -4.4] | -3.5 [-4.6 to -2.4]
  Change in waist circumference after 6 mo | -5.9 [-7.1 to -4.7] | -4.0 [-5.2 to -2.8]
  Change in waist circumference after 12 mo | -6.7 [-8.5 to -4.9] | -5.0 [-6.8 to -3.2]

5. Primary Outcome: Predicted Mean Differences in Total Cholesterol Level From Baseline by Assigned Dietary Group
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mmol/L
  Change of total cholesterol after 3 mo | -0.09 [-0.21 to 0.04] | 0.03 [-0.10 to 0.16]
  Change of total cholesterol after 6 mo | -0.04 [-0.16 to 0.07] | 0.03 [-0.09 to 0.15]
  Change of total cholesterol after 12 mo | 0.05 [-0.11 to 0.20] | 0.03 [-0.13 to 0.18]

6. Primary Outcome: Predicted Mean Differences in LDL Cholesterol Level From Baseline, by Assigned Dietary Group
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mmol/L
  Change in LDL cholesterol level after 3 mo | -0.02 [-0.14 to 0.10] | 0.05 [-0.06 to 0.18]
  Change in LDL cholesterol level after 6 mo | -0.04 [-0.15 to 0.06] | 0.02 [-0.08 to 0.13]
  Change in LDL cholesterol level after 12 mo | -0.08 [-0.24 to 0.08] | -0.05 [-0.20 to 0.11]

7. Primary Outcome: Predicted Mean Differences in HDL Cholesterol From Baseline, by Assigned Dietary Group
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mmol/L
  Change in HDL cholesterol level after 3 mo | 0.03 [-0.02 to 0.09] | -0.03 [-0.09 to 0.02]
  Change in HDL cholesterol level after 6 mo | 0.10 [0.05 to 0.15] | -0.00 [-0.05 to 0.05]
  Change in HDL cholesterol level after 12 mo | 0.24 [0.17 to 0.31] | 0.06 [-0.01 to 0.13]

8. Primary Outcome: Predicted Mean Differences in Total-HDL Cholesterol Ratio From Baseline, by Assigned Dietary Group
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
ratio
  Change in Total-HDL cholesterol ratio after 3 mo | -0.13 [-0.28 to 0.03] | 0.13 [-0.02 to 0.29]
  Change in Total-HDL cholesterol ratio after 6 mo | -0.25 [-0.38 to -0.11] | 0.07 [-0.06 to 0.21]
  Change in Total-HDL cholesterol level after 12 mo | -0.49 [-0.68 to -0.29] | -0.05 [-0.24 to 0.14]

9. Primary Outcome: Predicted Mean Differences in Triglycerides From Baseline, by Assigned Dietary Group
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mmol/L
  Change in Triglycerides after 3 mo | -0.21 [-0.32 to -0.11] | 0.03 [-0.08 to 0.14]
  Change in Triglycerides after 6 mo | -0.22 [-0.31 to -0.13] | -0.01 [-0.10 to 0.09]
  Change in Triglycerides after 12 mo | -0.23 [-0.34 to -0.12] | -0.07 [-0.18 to 0.04]

10. Primary Outcome: Predicted Mean Differences in Systolic Blood Pressure From Baseline, by Assigned Dietary Group
Description: as for outcome 4
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mm Hg
  Change in Systolic Blood Pressure after 3 mo | -4.2 [-5.9 to -2.5] | -2.6 [-4.3 to -0.9]
  Change in Systolic Blood Pressure after 6 mo | -2.9 [-4.5 to -1.3] | -2.2 [-3.8 to -0.6]
  Change in Systolic Blood Pressure after 12 mo | -0.2 [-2.6 to 2.1] | -1.3 [-3.6 to 1.0]

11. Primary Outcome: Predicted Mean Difference in Diastolic Blood Pressure, by Assigned Dietary Group
Description: Mean Difference in Diastolic Blood Pressure predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mm Hg
  Change in Diastolic Blood Pressure after 3 mo | -2.3 [-3.5 to -1.1] | -0.9 [-2.1 to 0.4]
  Change in Diastolic Blood Pressure after 6 mo | -1.7 [-2.8 to -0.5] | -0.5 [-1.7 to 0.6]
  Change in Diastolic Blood Pressure after 12 mo | -0.5 [-2.2 to 1.3] | 0.2 [-1.5 to 1.9]

12. Primary Outcome: Predicted Mean Difference in Plasma Glucose Level, by Assigned Dietary Group
Description: Mean Difference in Plasma Glucose Level predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mmol/L||
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
mmol/L||
  Change in Plasma Glucose Level after 3 months | -0.05 [-0.16 to 0.05] | -0.10 [-0.21 to 0.01]
  Change in Plasma Glucose Level after 6 months | 0.03 [-0.13 to 0.07] | -0.10 [-0.20 to 0.01]
  Change in Plasma Glucose Level after 12 months | 0.02 [-0.11 to 0.14] | -0.10 [-0.22 to 0.03]

13. Primary Outcome: Predicted Mean Differences in Serum Insulin Level From Baseline, by Assigned Dietary Group
Description: Mean Difference in Serum Insulin Level predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
pmol/L
  Change in Serum Insulin Level after 3 mo | -25.0 [-36.1 to -13.9] | -18.8 [-29.9 to -7.0]
  Change in Serum Insulin Level after 6 mo | -21.5 [-31.3 to -11.8] | -20.8 [-30.6 to -11.1]
  Change in Serum Insulin Level after 12 mo | -13.9 [-25.7 to -2.8] | -24.3 [-36.1 to -13.2]

14. Primary Outcome: Predicted Mean Differences in C-reactive Protein Level From Baseline, by Assigned Dietary Group
Description: Mean Difference in C-reactive Protein Level predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
nmol/L
  Change in Serum Creatinine Level after 3 mo | -4.8 [-13.3 to 3.8] | 5.7 [-2.9 to 13.3]
  Change in Serum Creatinine Level after 6 mo | -4.8 [-12.4 to 1.9] | 6.7 [-1.0 to 13.3]
  Change in Serum Creatinine Level after 12 mo | -6.7 [-16.2 to 2.9] | 8.6 [-1.0 to 18.1]

15. Primary Outcome: Predicted Mean Differences in Serum Creatinine Level From Baseline, by Assigned Dietary Group
Description: Mean Difference in Serum Creatinine Level predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: µmol/L¶
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
µmol/L¶
  hange in Serum Creatinine Level after 3 mo | -0.1 [-3.4 to 3.3] | 1.8 [-1.7 to 5.2]
  hange in Serum Creatinine Level after 6 mo | -3.1 [-6.1 to -0.2] | -1.7 [-4.7 to 1.3]
  hange in Serum Creatinine Level after 12 mo | -9.2 [-13.1 to -5.4] | -8.5 [-12.3 to -4.6]

16. Primary Outcome: Predicted Mean Differences of 10-y Framingham Risk Score From Baseline, by Assigned Dietary Group
Description: Mean Difference in 10-y Framingham Risk Score predicted from random-effects models that included diet, time, and diet-by-time interaction term. Markov-chain Monte Carlo techniques were used to impute missing values.
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: % risk of developing CVD in next 10 yrs
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Number analyzed (Participants) | 75 | 73
% risk of developing CVD in next 10 yrs
  Change in 10-Y Framingham Risk Score after 3 mo | -0.5 [-1.0 to 0.0] | 0.4 [-0.1 to 0.9]
  Change in 10-Y Framingham Risk Score after 6 mo | -0.7 [-1.0 to -0.3] | 0.4 [0.0 to 0.8]
  Change in 10-Y Framingham Risk Score after 12 mo | -1.0 [-1.6 to -0.5] | 0.4 [-0.2 to 0.9]

ADVERSE EVENTS:
Arm/Group | Low Carbohydrate Diet | Low Fat Diet
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/73
Other Adverse Events (participants affected / at risk) | 19/75 | 23/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Carbohydrate Diet (N=75) | Low Fat Diet (N=73)
Constipation at 3 months (Gastrointestinal disorders) | 19 | 13
Constipation at 6 months (Gastrointestinal disorders) | 18 | 19
Constipation at 12 months (Gastrointestinal disorders) | 1 | 17
Fatigue at 3 months (General disorders) | 17 | 9
Fatigue at 6 months (General disorders) | 18 | 22
Fatigue at 12 months (General disorders) | 15 | 16
Headache at 3 months (General disorders) | 6 | 18
Headache at 6 months (General disorders) | 12 | 16
Headache at 12 months (General disorders) | 11 | 22
Thirst at 3 months (General disorders) | 14 | 6
Thirst at 6 months (General disorders) | 12 | 9
Thirst at 12 months (General disorders) | 12 | 10
Polyuria at 3 months (General disorders) | 3 | 8
Polyuria at 6 months (General disorders) | 4 | 5
Polyuria at 12 months (General disorders) | 2 | 4
Diarrhea at 3 months (Gastrointestinal disorders) | 4 | 5
Diarrhea at 6 months (Gastrointestinal disorders) | 5 | 5
Diarrhea at 12 months (Gastrointestinal disorders) | 1 | 3
Heartburn at 3 months (Gastrointestinal disorders) | 7 | 12
Heartburn at 6 months (Gastrointestinal disorders) | 12 | 7
Heartburn at 12 months (Gastrointestinal disorders) | 9 | 18
Gas at 3 months (Gastrointestinal disorders) | 19 | 15
Gas at 6 months (Gastrointestinal disorders) | 17 | 22
Gas at 12 months (Gastrointestinal disorders) | 16 | 23
Nausea at 3 months (General disorders) | 4 | 2
Nausea at 6 months (General disorders) | 0 | 2
Nausea at 12 months (General disorders) | 0 | 3
Vomiting at 3 months (Gastrointestinal disorders) | 1 | 0
Vomiting at 6 months (Gastrointestinal disorders) | 0 | 0
Vomiting at 12 months (Gastrointestinal disorders) | 0 | 0
Decreased appetite (General disorders) | 3 | 1
Decreased appetite (General disorders) | 0 | 2
Decreased appetite (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes